CLINICAL TRIAL: NCT06045728
Title: Effect of Telerehabilitation on Overactive Bladder Symptoms and Metabolic Health in Obese Women
Brief Title: Telerehabilitation for Overactive Bladder Syndrome in Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Ibrahim Abdelmohsen Alghitany, teacher at Faculty of physical therapy Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004621
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Overactive Bladder Syndrome
MeSH Terms: interventions — Exercise Movement Techniques; Diet, Mediterranean

STUDY DESIGN:
Who Masked: Investigator
Masking Description: For insulin resistance the investigator will not know which group will be assessed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 telerehabilitation group (Active Comparator): subjects in this group will receive telerehabilitation sessions through online video programs (including Pilates exercise and diet) 3 times per week for 12 weeks. Outcome measures will be evaluated at baseline and after 12 weeks
  Interventions: Other: Pilates exercises; Behavioral: Mediterranean diet
- group 2 control group (Other): subjects in this group will be informed about the importance of Pilates exercise and diet for one session only. subjects will be asked to apply the exercise at home 3 times per week for 12 weeks and diet. Outcome measures will be evaluated at baseline and after 12 weeks
  Interventions: Other: Pilates exercises; Behavioral: Mediterranean diet

INTERVENTIONS:
Other: Pilates exercises — Pilates is a group of low impact muscle exercises that strengthen abdominal muscles, back, hips and pelvic floor muscles. the exercise consists of 10 min warm up, 40 min exercise and 10 min cooling down. the exercises that will be included: spine twist, double leg stretch, double leg circles, side leg circle, curl up, shoulder bridges and pelvic curl.
Behavioral: Mediterranean diet — it is a type of diet used for obesity management based on high vegetable intake, olive oil as a source of fat, the consumption of grains, legumes, and nuts with high amounts of pulp, low-medium consumption of fish, low consumption of red meat.

SUMMARY:
Overactive bladder syndrome(OAB) is a chronic medical condition which has a major influence on the quality of life in a significant amount of the population. The goal of this clinical trial study to identify the effect of telerehabilitation program on overactive bladder symptoms and metabolic health in obese women and to compare between the telerehabilitation group and the control group regarding overactive bladder symptoms and metabolic health in obese women.

DETAILED DESCRIPTION:
overactive bladder syndrome occurs globally and affects both genders with studies indicating high prevalence in obese females. Obesity brings with it not only an increased risk of cardiovascular diseases, but also urological dysfunction including overactive bladder. Pilates exercise and diet can be used as ways for controlling overactive bladder symptoms and improving overall health of obese subjects. Integration of telerehabilitation in the clinical practice benefits both providers and patients as well decreasing healthcare costs, so the objective of this study to determine the effect of telerehabilitation on overactive bladder symptoms and metabolic health in obese women through Pilates exercise and Mediterranean diet .

ELIGIBILITY:
Inclusion Criteria:

* women aged 35-45 years old
* class I obesity(30-34.9kg/m2)
* women will be referred by urologist with Presence of overactive bladder symptoms confirmed by overactive bladder questionnaire
* waist circumference more than 88 cm

Exclusion Criteria:

* history of surgical treatment of urological disease
* infection of urinary tract
* oncological and neurological urinary tract disease,
* refusal to participate in the study

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — because prevalence of overactive bladder symptoms in obese women is high
Enrollment: 80 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
body mass index | at baseline and after 12 weeks of the intervention
  it is calculated by dividing weight in kg on height in m square
waist circumference | at baseline and after 12 weeks of the intervention
  it is an indicator of central obesity with waist circumference more than 88 cm is considered central obesity in females
overactive bladder questionnaire short form | at baseline and after 12 weeks of the intervention
  is a questionnaire that is divided into two sections : symptoms and quality of life. In symptoms section, the higher the scores the more the symptoms that bother the patients. higher scores in quality of life section indicates better quality of life.
patient perception of intensity of urgency scale | at baseline and after 12 weeks of the intervention
  a scale ranges from 0 to 4 that measures the degree of urgency with micturition with higher scores indicate higher perception of urgency
HOMA IR | at baseline and after 12 weeks of the intervention
  The homeostatic model assessment (HOMA IR) is a method used to quantify insulin resistance . derived from the product of the insulin and glucose values divided by a constant.

SECONDARY OUTCOMES:
telehealth usability questionnaire | after 12 weeks of the intervention
  a comprehensive questionnaire that covers all usability factors (i.e., usefulness, ease of use, effectiveness, reliability, and satisfaction). It is used with various types of telehealth systems, including the traditional videoconferencing systems, computer-based systems, and the mobile telehealth systems.

CONTACTS AND LOCATIONS:
Overall Officials: salma I alghitany, PHD, Study Director — Cairo University
Locations (1):
- Online Video Programs With Patients Referred From Urologist ( Kasr Eleiny Hospital), Giza, Egypt

REFERENCES:
- See also: Relationship Between Central Obesity, General Obesity, Overactive Bladder Syndrome and Urinary Incontinence Among Male and Female Patients Seeking Care for Their Lower Urinary Tract Symptoms — https://doi.org/10.1016/j.urology.2018.09.012